CLINICAL TRIAL: NCT04534192
Title: Physician Initiated, Prospective, Non-randomized Single-centre, Single-arm Trial, Investigating the Safety and Efficacy of the Treatment With the Non-compliant Jade Balloon in TASC C and D Athero-occlusive Infra-inguinal Disease in Patients With Chronic Limb Threatening Limb Ischemia From SingaporE (PINNACLE)
Brief Title: Investigating the Safety and Efficacy of the Treatment With the Non-compliant Jade Balloon in TASC C and D Athero-occlusive Infra-inguinal Disease in Patients With Chronic Limb Threatening Limb Ischemia From SingaporE
Acronym: PINNACLE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Singapore General Hospital (Other)
Collaborators: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020/2425
Record Dates: First submitted 2020-08-26; First posted 2020-09-01 (Actual); Last update posted 2020-11-02 (Actual); Status verified 2020-10

CONDITIONS: Critical Limb Ischemia; Peripheral Artery Disease
Keywords: non-compliant high pressure balloon; JADE
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia; Peripheral Arterial Disease

STUDY DESIGN:
Intervention Model Description: Non-randomized, single arm
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- JADE balloon (Experimental): Non-compliant high pressure JADE balloon for the treatment of infrainguinal stenotic occlusive or stenotic TASC C & D lesions in patients with chronic limb threatening ischemia.
  Interventions: Device: JADE Balloon

INTERVENTIONS:
Device: JADE Balloon — Suitable TASC C and D lesions will be treated with non-compliant high pressure JADE balloon.

SUMMARY:
The objective of this clinical study is to evaluate the 6-month safety and performance outcome of the non-compliant high pressure JADE balloon for the treatment of infrainguinal stenotic occlusive or stenotic TASC C & D lesions in patients with chronic limb threatening ischemia.

DETAILED DESCRIPTION:
Pulsatile straight line blood flow to the foot is required to aid wound healing in the setting of chronic limb threatening ischaemia (CLTI). Patients with CLTI usually present with infra-popliteal arterial occlusions and endovascular therapies to restore blood flow are often preferred considering their inherently less invasive nature and because of multiple patient background comorbidities or absence of a suitable vein conduit in these patients. Below The Knee (BTK) plain balloon angioplasty (POBA) remains the only viable "standard of care" in the management of long "Real World" BTK Lesions. However tibial angioplasty is plagued by high rate of re-occlusion/stenosis because of barotrauma caused by the intra-arterial ballooning and subsequent development of neointimal hyperplasia. Devices coated with paclitaxel have been used successfully to limit restenosis by inhibiting the biologic pathway that leads to intimal hyperplasia. However, a recent formal systematic review and study-level meta-analysis of randomized controlled trials investigating treatment of the infra-popliteal arteries with paclitaxel-coated balloons compared with conventional balloon angioplasty for critical limb ischemia (CLI) was recently published showing amputation-free survival was significantly worse in use of paclitaxel coated balloons compared to plain angioplasty. Furthermore current poor patency seen in BTK angioplasty is likely contributed in part by small vessel size and poor luminal gain after standard semi-compliant POBA. Vessel Preparation and Optimising POBA with High Pressure, Non-Compliant balloons may help achieve Luminal Gain for rapid and sustained flow for wound healing. The objective of this clinical study is to evaluate the 6-month safety and performance outcome of the non-compliant high pressure JADE balloon for the treatment of infrainguinal stenotic occlusive or stenotic TASC C & D lesions in patients with chronic limb threatening ischemia.

ELIGIBILITY:
Inclusion Criteria:

1. Age of subject is > 40 years old. Patient covered by MediShield insurance as provided by Singapore government.
2. Patient has critical limb ischemia, presenting a score from 4 to 6 following the Rutherford classification
3. Patients must agree to return for all required post-index procedure follow-up visits.
4. Patient understands the nature of the procedure and provides written informed consent, prior to enrolment in the study
5. Patient has a projected life expectancy of at least 12 months and has not suffered a myocardial infarction within past 30 days

Angiographic Inclusion Criteria:

1. De novo and post-PTA re-stenotic lesions located in the superficial femoral, popliteal and tibial arteries suitable for endovascular therapy
2. The target lesion is located within the native SFA/popliteal/tibial artery
3. The length of the target lesion(s) is > 100mm and considered as TASC C or D lesion according to the TASC II classification.
4. The target lesion has angiographic evidence of stenosis > 50% or occlusion, which has been passed with standard guidewire manipulation and no other adjunctive devices have been used to prepare the lesion (example scoring balloon, rotablator, atherectomy device)
5. Target vessel diameter visually estimated is >1.5mm and < 6.5mm below the groin
6. Prior to enrolment, the guidewire has crossed the target lesion
7. Lesions in the treated segment may be continuous or may have gaps present between stenoses and occlusions
8. Inflow iliac, common femoral artery lesions can be treated during the same procedure using standard angioplasty and/or approved device/open surgery. These inflow lesions must be treated first prior to consideration of treatment of the distal lying lesions. The patient can be enrolled if the inflow lesions are treated with good embolization)
9. There is angiographic evidence of at least one- vessel-runoff through the ankle and into the foot, irrespective of whether or not outflow was re- established by means of previous endovascular intervention

Exclusion Criteria:

1. Patient is permanently wheel-chair bound or bedridden
2. Presence of a stent in the target lesion(s) that was placed during a previous procedure
3. The intervention is being performed in preparation for a planned amputation.
4. Untreated flow-limiting inflow lesions
5. Any previous surgery in the target vessel (including prior ipsilateral crural bypass)
6. Previous bypass surgery in the same limb
7. Patients with a history of Myocardial Infarction (MI), thrombolysis or angina within 30 days prior-index procedure.
8. Patients with a history of major disabling stroke within 3 months prior index procedure.
9. Patients with any type of previous or planned surgical or interventional procedure within 15 days prior- and/or within 30 days post-index procedure.
10. Untreatable lesion located at the distal outflow arteries
11. Patients with uncorrected bleeding disorders
12. Aneurysm located at the level of the SFA/popliteal artery
13. Non-atherosclerotic disease resulting in occlusion (e.g. embolism, Buerger's disease, vasculitis)
14. Any condition which prevents patient from complying with the study protocol or if patient has a life expectancy of <1yr.
15. Major distal amputation (above the transmetatarsal) in the study limb or non-study limb
16. Patients with a presence or history of severe renal failure (Glomerular Filtration Rate (GFR) ≤ 30 ml/min) and is not dialysis dependent.
17. Neurotrophic ulcer or heel pressure ulcer or ulcer potentially involving calcaneus (index limb)
18. Episode of acute limb ischaemia within the previous 1 month
19. Use of thrombectomy, cutting balloon, lithotripsy, atherectomy or laser devices during procedure
20. Any patient considered to be hemodynamically unstable at onset of procedure
21. Patients with a known hypersensitivity or contraindication to aspirin, heparin, clopidogrel, or other anticoagulant/anti-platelet therapies or sensitivity to contrast media that cannot be adequately premedicated.
22. The patient is currently breast-feeding, pregnant or intends to become pregnant.
23. Subject receiving immunosuppression therapy, or has known serious immunosuppressive disease (e.g., human immunodeficiency virus), or has severe autoimmune disease that requires chronic immunosuppressive therapy (e.g., systemic lupus erythematosus, etc.) The patient should also not receive inhibitors of CYP3A (such as Itraconazole, and Erythromycin), or inducers of CYP3A (such as Rifampin) within 90 days following the procedure.
24. Patient is participating in another research study of a device, medication, biologic or other agent within 30 days which could in the opinion of the investigator affect the results of this study
25. Patients with any contraindications as mentioned in the Instructions for Use (IFU) of the Investigational Device.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2022-03-01 (Estimated); Study Completion 2022-08-01 (Estimated)

PRIMARY OUTCOMES:
Freedom from Major Adverse Events | 30 days post-index procedure
  A composite of freedom from device- and procedure-related mortality through 30 days
Performance Primary Endpoint | 6 months post-index procedure
  Freedom from clinically driven target lesion revascularization (TLR) within 6 months post-index procedure. (Clinically driven TLR is defined as any re-intervention performed for ≥ 50% diameter stenosis (visual estimate) at the target lesion after documentation of recurrent or unresolved and continuing clinical symptoms of the patient.)

SECONDARY OUTCOMES:
Primary patency rate | 6- and 12-month post-index procedure
  defined as absence of a hemodynamically significant stenosis on Duplex ultrasound (systolic velocity ratio no greater than 2.5) at the target lesion and without TLR within the time of procedure and the given follow-up. Note: Any patient where DUS is not analysable at index and/or at follow-up, where there is documented significant progression of disease above the target lesion, or who undergo a major amputation prior to the time of follow-up will be excluded from the calculation of this endpoint.
Technical success | Immediately post-op
  defined as the ability to cross and dilate the lesion and achieve residual angiographic stenosis no greater than 30%
Freedom from clinically-driven TLR | 12-month post-index procedure
  defined as a repeat intervention to maintain or re-establish patency within the region of the treated arterial vessel plus 5mm proximal and distal to the treated lesion edge at the respective time points
Clinical success at follow-up | 6 and 12 months post index procedure
  defined as an improvement of Rutherford classification at all follow- up time points of one class or more as compared to the pre-procedure Rutherford classification
Wound healing | 6 months post-index procedure
  closure of primary wound by more than 70%
Freedom from major target limb amputation (above ankle) | 6 months and 12 months post-index procedure
Improvements in walking | 3, 6 and 12 months post-index procedure.
  Comparison of the scores on the Walking Impairment Questionnaire (WIQ) between baseline and follow-ups.
Freedom from serious adverse events | 3, 6 and 12 months post-index procedure.
  as defined per ISO 14155:2011

CONTACTS AND LOCATIONS:
Overall Officials: Tjun Yip Tang, MD, Principal Investigator — Singapore General Hospital
Locations (1):
- Singapore General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No